CLINICAL TRIAL: NCT03908944
Title: Postoperative Pain and Headache After Craniotomy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI- Dr. Jellish passed away. The study was terminated with the IRB
Sponsor: Steven Edelstein (Other)
Responsible Party: Sponsor-Investigator, Steven Edelstein, Anesthesiology, Vice-Chairman, Loyola University
Organization: Loyola University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 210979
Record Dates: First submitted 2019-03-29; First posted 2019-04-09 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Methadone; Standard of Care

STUDY DESIGN:
Who Masked: Participant
Masking Description: Study participant will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard of Care (Active Comparator): Standard of Care patients will be given an infusion of remifentanil 0.15-0.25 mcg/kg/min as part of their intraoperative anesthetic regimen. The infusion will be maintained until the end of surgery and will be discontinued upon emergence. Prior to emergence, 100-200 mcg of fentanyl will be titrated for additional analgesia after emergence.
  Interventions: Drug: Standard of Care
- Methadone (Experimental): Individuals in this group will receive an identical anesthetic without the addition of remifentanil. They will be given methadone 0.2 mg/kg IV at the beginning of the anesthetic. A lidocaine bolus of 1.5 mg/kg will be given with induction of anesthesia followed by an infusion of lidocaine at 2 mg/kg/hr until the end of surgery.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — Individuals in this group will receive an identical anesthetic without the addition of remifentanil. They will be given methadone 0.2 mg/kg IV at the beginning of the anesthetic. A lidocaine bolus of 1.5 mg/kg will be given with induction of anesthesia followed by an infusion of lidocaine at 2 mg/kg/hr until the end of surgery.
  Arms: Methadone
Drug: Standard of Care — Standard of Care patients will be given an infusion of remifentanil 0.15-0.25 mcg/kg/min as part of their intraoperative anesthetic regimen. The infusion will be maintained until the end of surgery and will be discontinued upon emergence. Prior to emergence, 100-200 mcg of fentanyl will be titrated for additional analgesia after emergence.
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to assess the outcomes of an anesthetic technique which is not synthetic opioid based, on postoperative pain modulation and development of post craniotomy headache against a cohort of patients where an opioid based standard anesthetic technique was used for craniotomy. The hypothesis that is tested is that the use of agents other than synthetic short acting opioids will reduce the amount of postoperative pain and the incidence of headache after surgery.

DETAILED DESCRIPTION:
120 ASA physical status I to III patients, ages 18 to 75, who are to undergo supratentorial, infratentorial or skull base tumor resection will be included in this randomized control study. The Preadmission Testing is done for the most part in the same day the patient has an ENT clinic appointment or just Anesthesia preadmission screening date. This is the day that patient will come to the clinic for pre-admission testing, days before the plan procedure. They will meet with Anesthesiology department clinician. Having the consent process started in the preadmission Clinic with Anesthesiology clinician will be better for the patient to process and understand the information about the study before agreeing to participate. If the patient is only coming In the ENT Clinic then the patient will be approached about the study in the ENT clinic. At the day of the surgery if the patent have any additional question or any unclear information, the PI or the Co-PI will answer before the patient signing the consent. Patients who are pregnant, undergoing emergency, neurovascular, or trigeminal nerve pain procedures, those unable to give informed consent, or who were extremely debilitated (ASA physical status IV or V) in liver or renal failure will be excluded from the study. A mini mental status exam will be performed on the day of surgery before the patient presents to the operating room. All patients will receive a general anesthetic consisting of propofol 2 mg/kg intravenously (IV) and fentanyl 2 mcg/kg IV induction of anesthesia followed by maintenance anesthetic consisting of desflurane 5% to 6% end tidal concentration. All patients will be given rocuronium 0.1 mg/kg/IV or succinylcholine 1.0 mg/kg IV to facilitate intubation along with a 70/30 mixture of air in 02. Patients will be assigned via a computer generated randomization table before surgery to receive one of two anesthetic techniques perioperatively.

Group 1 patients will be given an infusion of remifentanil 0.15-0.25 mcg/kg/min as part of their intraoperative anesthetic regimen. The infusion will be maintained until the end of surgery and will be discontinued upon emergence. Prior to emergence, 100-200 mcg of fentanyl will be titrated for additional analgesia after emergence.

Group 2 individuals will receive an identical anesthetic without the addition of remifentanil.. They will also be given methadone 0.2 mg/kg IV at the beginning of the anesthetic. A lidocaine bolus of 1.5 mg/kg will be given with induction of anesthesia followed by an infusion of lidocaine at 2 mg/kg/hr until the end of surgery.

ELIGIBILITY:
Patient Inclusion Criteria:

* Undergoing Supratentorial, Infratentorial or Skull Base Tumor resection.
* Age 18 to 75
* ASA physical status I to III

Patient Exclusion Criteria:

* ASA physical status IV or V
* Allergies to the medication used for the study
* Pregnant
* Undergoing Emergency, Neurovascular, or Trigeminal Nerve pain procedure
* Liver or renal failure
* Unable to give informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2021-01-02 (Estimated); Study Completion 2022-01-02 (Estimated)

PRIMARY OUTCOMES:
Post craniotomy pain | 6 months
  Assessed via a Verbal Analog Scale from 0-10 with 0 being no pain and 10 being the worst pain ever experienced
Headache intensity | 6 months
  Assessed via qualitative rating of sharp, dull, pressure, or incisional pain

CONTACTS AND LOCATIONS:
Overall Officials: Walter Jellish, MD/Ph.D, Principal Investigator — Loyola University; Steven Edelstein, MD, Study Director — Loyola University
Locations (1):
- Loyola Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share individual Data.

REFERENCES:
- [Background] De Benedittis G, Lorenzetti A, Migliore M, Spagnoli D, Tiberio F, Villani RM. Postoperative pain in neurosurgery: a pilot study in brain surgery. Neurosurgery. 1996 Mar;38(3):466-9; discussion 469-70. doi: 10.1097/00006123-199603000-00008. PMID 8837797
- [Background] de Gray LC, Matta BF. Acute and chronic pain following craniotomy: a review. Anaesthesia. 2005 Jul;60(7):693-704. doi: 10.1111/j.1365-2044.2005.03997.x. PMID 15960721
- [Background] Mosek AC, Dodick DW, Ebersold MJ, Swanson JW. Headache after resection of acoustic neuroma. Headache. 1999 Feb;39(2):89-94. doi: 10.1046/j.1526-4610.1999.3902089.x. PMID 15613200
- [Background] Koperer H, Deinsberger W, Jodicke A, Boker DK. Postoperative headache after the lateral suboccipital approach: craniotomy versus craniectomy. Minim Invasive Neurosurg. 1999 Dec;42(4):175-8. doi: 10.1055/s-2008-1053393. PMID 10667820
- [Background] Pedrosa CA, Ahern DK, McKenna MJ, Ojemann RG, Acquadro MA. Determinants and impact of headache after acoustic neuroma surgery. Am J Otol. 1994 Nov;15(6):793-7. PMID 8572094
- [Background] Vijayan N. Postoperative headache in acoustic neuroma. Headache. 1995 Feb;35(2):98-100. doi: 10.1111/j.1526-4610.1995.hed3502098.x. PMID 7737870
- [Background] Lai J, Porreca F, Hunter JC, Gold MS. Voltage-gated sodium channels and hyperalgesia. Annu Rev Pharmacol Toxicol. 2004;44:371-97. doi: 10.1146/annurev.pharmtox.44.101802.121627. PMID 14744251
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Jellish WS, Leonetti JP, Sawicki K, Anderson D, Origitano TC. Morphine/ondansetron PCA for postoperative pain, nausea, and vomiting after skull base surgery. Otolaryngol Head Neck Surg. 2006 Aug;135(2):175-81. doi: 10.1016/j.otohns.2006.02.027. PMID 16890064
- [Background] Hawthorne G, Sansoni J, Hayes L, Marosszeky N, Sansoni E. Measuring patient satisfaction with health care treatment using the Short Assessment of Patient Satisfaction measure delivered superior and robust satisfaction estimates. J Clin Epidemiol. 2014 May;67(5):527-37. doi: 10.1016/j.jclinepi.2013.12.010. PMID 24698296